CLINICAL TRIAL: NCT00322322
Title: Early Administration of L-carnitine in Hemodialysis Patients: Double Blind Randomized Trial Versus Placebo
Brief Title: Early Administration of L-carnitine in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle BRINDEL, Department of Clinical Research of developpement
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P050316
Record Dates: First submitted 2006-05-03; First posted 2006-05-05 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2007-03

CONDITIONS: Complication of Hemodialysis; Hyperthyroidism Treated or Under Control
Keywords: L-carnitine supplementation; Hemodialysis; Anaemia; Erythropoietin responsiveness
MeSH Terms: conditions — Anemia | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): L-Carnitine
  Interventions: Drug: L-Carnitine

INTERVENTIONS:
Drug: L-Carnitine — L-Carnitine

SUMMARY:
Hemodialysis is a cause of carnitine deficiency. The deficiency of carnitine induces an anemia by an increase fragility of the red blood cells, a muscular fatigue and a cardiac dysfunction. We proposed to evaluate the benefit of an early administration of L-carnitine in hemodialysis patients. The patients should be included in the first month after the start of chronic hemodialysis, randomized to receive L-carnitine or placebo and should be followed-up during one year.

DETAILED DESCRIPTION:
The first aim of the study is to compare the resistance index to erythropoietin (hemoglobin level / rHuerythropoietin dose) with L-carnitine versus placebo Double blind randomized study evaluating the supplementation with L-carnitine versus placebo in patients beginning chronic hemodialysis for less than 1 month.

Primary outcome to compare rHuerythropoietin resistance index defined as hemoglobin level / rHuEPO dose ratio with L-carnitine and with placebo.

Secondary endpoints to compare acylcarnitine / carnitine ratio, number of red blood cells transfusion, physical status, quality of life, hypotensive episodes, lipid profile, diabetes profile, albuminemia, c reactive protein.

Several variables that influenced primary and secondary endpoints will be included in a multivariate analysis; albuminemia, c reactive protein, iron status, dialysis efficiency, protein intake, lipid intake, treatment with additional vitamins (C, B9, B6), treatment with statins, treatment of predialysis hypotension by midodrine, antihypertensive treatments.

Statistical analysis:

* description of the cohort
* comparisons of each evaluated variables between the 2 treatments
* ANOVA study for repeated measurements from inclusion to month-12 for Hb / rHuEPO dose to compare the course of the ratio between each group in intention to treat analysis
* analysis of the ratio Hb / rHuEPO month by month and taking into account tempera withdrawal

Following analysis in both intention to treat and per protocol analysis:

* acylcarnitine / carnitine ratio by ANOVA for repeated data
* number of predialysis hypotension by Chi2 test
* number of red blood cells transfusion by Chi2 test
* SF-36 physical status by comparison of mean
* SF-36 total score by comparison of mean
* lipid profile by ANOVA for repeated data
* HbA1c by ANOVA for repeated data
* variables that influenced primary and secondary variables will be analyzed by multivariate analysis
* statistical study of clinical events per month

ELIGIBILITY:
Inclusion Criteria:

* Patient with less than 1 month on hemodialysis.
* Treated with rHuEPO.
* Male or female aged of more than 18 years old.
* With contraception treatment for women of procreation age.
* Having received and understand information.

Exclusion Criteria:

* Patients with no need of rHuEPO
* Patients with cancer disease
* Patients with life expectancy under 6 months
* Patients having a proved carnitine deficiency before the start of hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Resistance index to erythropoietin | during de study
  Resistance index to erythropoietin
Haemoglobin level/weekly rHuerythropoietin dose in patients receiving l-carnitine versus those receiving the placebo. | during the study
  Haemoglobin level/weekly rHuerythropoietin dose in patients receiving l-carnitine versus those receiving the placebo.

SECONDARY OUTCOMES:
Acylcarnitine/carnitine ratio measured quarterly | during the study
  Acylcarnitine/carnitine ratio measured quarterly
Number of red blood cells transfusion per patient during the study, data collected monthly | during the study
  Number of red blood cells transfusion per patient during the study, data collected monthly
Predialysis hypotension per patient during the study, data collected monthly | during the study
  Predialysis hypotension per patient during the study, data collected monthly
SF 36 physical and total score at inclusion and at the end of the study | during the study
  SF 36 physical and total score at inclusion and at the end of the study
Lipid profile, measured quarterly | during the study
  Lipid profile, measured quarterly
HbA1c, measured quarterly for diabetic patients and patients with glucose intolerance | during the study
  HbA1c, measured quarterly for diabetic patients and patients with glucose intolerance
Albuminemia measured quarterly | during the study
  Albuminemia measured quarterly
c reactive protein measured quarterly | during the study
  c reactive protein measured quarterly

CONTACTS AND LOCATIONS:
Overall Officials: Lucile Mercadal, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Assistance Publique Hopitaux de Paris, Paris
  - HOPITAL LA PITIE SALPETRIERE, service de Néphrologie, Paris

REFERENCES:
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822
- [Derived] Nishioka N, Luo Y, Taniguchi T, Ohnishi T, Kimachi M, Ng RC, Watanabe N. Carnitine supplements for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013601. doi: 10.1002/14651858.CD013601.pub2. PMID 36472884
- [Derived] Mercadal L, Tezenas du Montcel S, Chonchol MB, Debure A, Depreneuf H, Servais A, Bassilios N, Assogba U, Allouache M, Prie D. Effects of L-Carnitine on Mineral Metabolism in the Multicentre, Randomized, Double Blind, Placebo-Controlled CARNIDIAL Trial. Am J Nephrol. 2018;48(5):349-356. doi: 10.1159/000494338. Epub 2018 Nov 8. PMID 30408788